CLINICAL TRIAL: NCT00843037
Title: A Investigator Initiated Phase II Study Of Sunitinib In Patients With Recurrent Paraganglioma/Pheochromocytoma
Brief Title: Study Of Sunitinib In Patients With Recurrent Paraganglioma/Pheochromocytoma
Acronym: SNIPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNIPP
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Paraganglioma; Pheochromocytoma
Keywords: PARAGANGLIOMA; PHEOCHROMOCYTOMA; SUNITINIB; PHASE II; Metastatic or locally advanced malignant paraganglioma; Metastatic or locally advanced malignant pheochromocytoma
MeSH Terms: conditions — Paraganglioma; Pheochromocytoma; Neoplasm Metastasis | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label - Sunitinib (Experimental): Sunitinib, 50mg daily, once daily for 4 weeks followed by a 2-week break
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 50 mg oral dose daily for 4 weeks, 2 week rest period (repeating 6 week cycles)
  Other Names: Sunitinib malate (suntinib; SU11248, SU011248, Sutent®)

SUMMARY:
This is an open-label phase II study of an investigational drug, sunitinib malate in patients with advanced malignant paraganglioma or phaeochromocytoma cancer. Paragangliomas (PGs) are tumours that arise from the para-sympathetic system in the head and neck and sympathetic system in the thorax and abdomen. Paragangliomas that secrete hormones (catecholamines) from the adrenal glands are called pheochromocytomas (PCs). In this study, patients whose disease has advanced or spread despite prior standard therapy, will receive sunitinib for 4-weeks followed by a 2-week rest period, for up to 12 months, in the absence of disease progression. Sunitinib is an investigational drug, which has been shown to shrink tumours in several tumour models. The study will evaluate the efficacy as well as the toxicity profile of sunitinib when used as an alternative treatment for patients with PG/PC tumours.

DETAILED DESCRIPTION:
This study will be a single arm, open-label, phase II trial of sunitinib in patients with metastatic or locally advanced malignant paraganglioma or phaeochromocytoma. Oral sunitinib (50 mg) will be administered to all patients daily for the first four weeks of a six week study cycle, followed by a 2-week rest. Patients will be assessed for response to study treatment using MRI/CT scans as well as bio-chemical tests, and will receive the study treatment for up to 12 months or until disease progression.

Primary study outcomes include:

To assess the efficacy (response rate) of sunitinib given orally daily for 4 out of every 6 weeks in patients with advanced or metastatic paraganglioma/ pheochromocytoma.

To assess the toxicity of sunitinib in patients with advanced or metastatic paraganglioma/ pheochromocytoma.

To document effects of sunitinib on markers of biochemical activity of advanced or metastatic paraganglioma/ pheochromocytoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of malignant paraganglioma or pheochromocytoma and either evidence of metastases or unresectability.
* Evidence of recent disease progression (radiological, biochemical, symptomatic).
* Measurable disease defined as that which can be measured in at least one dimension with a minimum size of 10 mm by CT scan.
* ECOG 0-2.
* Life expectancy of greater than 24 weeks.
* Age > 18 years.
* Patients must have normal organ and marrow function.
* Patients must have PT/INR/PTT within 1.2 X the upper limit
* Patients may have had prior radiation therapy. A minimum of 28 days must have elapsed between the end of radiotherapy and registration onto the study.
* Previous Surgery: Previous major surgery is permitted provided that it has been at least 28 days prior to patient registration
* Laboratory Requirements Parameter Limit granulocytes (AGC) > 1.5 x 109/L platelets > 100 x 109/L bilirubin < 1.5XULN AST and ALT < 2.5 x ULN Amylase <1.5XULN Lipase <1.5XULN Calcium < 3 mmol/L creatinine < 2.0XULN

Exclusion Criteria:

* History of other malignancies.
* Patients with known brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib.
* Patients receiving concurrent treatment with other anti-cancer therapy given for paraganglioma or pheochromocytoma or other therapy or other investigational anticancer agents.
* Patients who have received prior treatment with any other antiangiogenic agent or multi-targeted tyrosine kinase inhibitors are ineligible.
* Patients with any of the following cardiovascular findings are to be excluded:
* QTc prolongation or other significant ECG abnormalities.
* Current or history of Class III or IV heart failure as defined by the NYHA functional classification system
* Patients with prior anthracycline exposure, previous central thoracic radiation that included heart in radiation port, or a history of NYHA Class II cardiac function.
* Poorly controlled hypertension
* Myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
* History of venous thrombosis or pulmonary embolism in the past 3 months
* History of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin
* Patients with bowel obstruction or any condition that impairs their ability to swallow and retain sunitinib tablets.
* Use of agents with proarrhythmic potential is not permitted during the study.
* Must be able to stop prohibited selected CYP3A4 inhibitors/inducers prior to starting sunitinib
* Patients with pre-existing hypothyroidism prior to enrolment are ineligible unless they are euthyroid on medication.
* Pregnant or lactating women, positive pregnancy test, women of childbearing potential who do not agree to use adequate contraception prior to study entry and for the duration of study participation.
* Known HIV-positive patients on combination antiretroviral therapy
* Greater than +1 proteinuria on urinary dipstick if also >1g urinary protein/24hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, MD, FRCPC, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (4):
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario
  - Hôpital Notre-Dame du CHUM, Montreal, Quebec
- University Medical Centre Groningen, Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between May 2009 and May 2016 from three centres within Canada and one in the Netherlands.
Pre-assignment Details: 25 of the planned 28 patients were enrolled
Groups:
- Single-Arm, Open Label - Sunitinib: Sunitinib: 50 mg oral dose daily for 4 weeks, 2 week rest period (repeating 6 week cycles)
Period: Overall Study
Arm/Group | Single-Arm, Open Label - Sunitinib
Started | 25
Completed | 24
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single-Arm, Open Label - Sunitinib
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 50 [17 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Canada | 24
  Netherlands | 1
Histology [Count of Participants; unit: Participants]
  Paraganglionoma | 11
  Pheochromocytoma | 14
Prior Systemic Therapy [Count of Participants; unit: Participants]
  Systemic adjuvant | 1
  Systemic advanced | 3
  None | 21
Prior Local Therapy [Count of Participants; unit: Participants]
  Radiation only | 4
  Surgery only | 11
  Surgery and radiation | 5
  None | 5
Stage [Count of Participants; unit: Participants]
  Metastatic | 23
  Locally advanced | 2
Sites of Mestastases [Number; unit: participants]
  Lymph Nodes | 11
  Lung | 12
  Bone | 12
  Liver | 14
Total Baseline Urine Metanephrines Elevated [Count of Participants; unit: Participants]
  Yes | 15
  No | 6
  Missing | 4
Reason for Enrollment [Count of Participants; unit: Participants]
  Radiologic and/or biochemical PD | 20
  Symptomatic PD | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) Which is Defined as Either a Partial Response (PR) Complete Response (CR) or Stable Disease (SD) for ≥ 12 Weeks Measured Using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria.
Description: The primary endpoint of this study was disease control rate (DCR) defined as a partial response (PR), complete response (CR), or stable disease maintained for ≥12 weeks from the initiation of treatment. Tumour response to sunitinib was assessed as per RECIST 1.1 using CT-imaging. Clinically apparent lesions needed to be >10mm by calliper measurement to be included as targets. The primary endpoint was met despite closing to accrual early.
Time Frame: Every 12 weeks (2 cycles) up to disease progression or study discontinuation (an average of 13.5 6-week cycles or about 1.5 years).
Population: Twenty-three patients were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open Label - Sunitinib
Number analyzed (Participants) | 23
Participants
  CR, PR, SD > 12 weeks | 19
  Not CR, PR, SD > 12 weeks | 4

2. Secondary Outcome: Biochemical Response (BCR) of > 20% Drop in 24-hour Urinary Metanephrines, Catecholamines or Serum Chromogranin A, Sustained for > 12-week Period
Description: Biochemical and symptom changes: timed urinary catecholamine collection over 24 h included measurements of norepinephrine, epinephrine, dopamine and total metanephrines.
Time Frame: Within 7 days of study registration and every 12 weeks (2 cycles) up to treatment discontinuation (an average of 13.5 6-week cycles or about 1.5 years).
Population: Includes patients that had F/U measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open Label - Sunitinib
Number analyzed (Participants) | 16
Participants
  24-h urinary metanephrines: number analyzed (Participants) | 12
  24-h urinary metanephrines: BCR >20% decline in values > 12 weeks | 7
  24-h urinary metanephrines: No BCR >20% decline in values > 12 weeks | 5
  norepinephrine: number analyzed (Participants) | 12
  norepinephrine: BCR >20% decline in values > 12 weeks | 7
  norepinephrine: No BCR >20% decline in values > 12 weeks | 5
  Epinephrine: number analyzed (Participants) | 5
  Epinephrine: BCR >20% decline in values > 12 weeks | 4
  Epinephrine: No BCR >20% decline in values > 12 weeks | 1
  Dopamine: number analyzed (Participants) | 5
  Dopamine: BCR >20% decline in values > 12 weeks | 3
  Dopamine: No BCR >20% decline in values > 12 weeks | 2
  Catecholamines (all): BCR >20% decline in values > 12 weeks | 11
  Catecholamines (all): No BCR >20% decline in values > 12 weeks | 5

3. Secondary Outcome: Overall Survival
Description: The median overall survival
Time Frame: From time of enrollment until loss to follow-up or death (approximately 125 months for longest patient on treatment).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single-Arm, Open Label - Sunitinib
Number analyzed (Participants) | 25
months | 112 [25.8 to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Time to Progression
Description: Median Progression-Free Survival (PFS)
Time Frame: as for outcome 1
Population: Includes patients that had a PFS event (up to 31 Jan 2018).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single-Arm, Open Label - Sunitinib
Number analyzed (Participants) | 21
months | 13.4 [5.3 to 24.6]

5. Secondary Outcome: Overall Response Rate (PR) + (CR)
Description: Overall response rate (PR) + (CR) of participants
Time Frame: as for outcome 1
Population: 23 evaluable for response data
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open Label - Sunitinib
Number analyzed (Participants) | 23
Participants
  CR+PR | 3
  Not CR or PR | 20

ADVERSE EVENTS:
Time Frame: From time of enrollment to 28 days post-discontinuation of treatment, with ongoing protocol-related toxicities and late toxicities followed until loss to follow-up or death (approximately 125 months for longest patient on treatment).
Arm/Group | Single-Arm, Open Label - Sunitinib
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Arm, Open Label - Sunitinib (N=25)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (3)
Death due to Progressive Disease (General disorders) | 2 (2)
Decompensated Heart Failure (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Elevated Creatinine/Renal failure (Renal and urinary disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Generalized Edema (General disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Hypertension crisis (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension and Electrolyte disorder (Vascular disorders) | 1 (1)
Ileus secondary to adherence (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC - urinary tract (Infections and infestations) | 1 (1)
Left Renal Vein Thrombosis (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Pulmonary Emboli (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Renal Colic (Renal and urinary disorders) | 1 (1)
Tachycardia, Palpitations (Cardiac disorders) | 1 (1)
Uncontrolled Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper GI Toxicity Post Radiotherapy (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Arm, Open Label - Sunitinib (N=25)
Fatigue (General disorders) | 17 (48)
Nausea/Vomiting (Gastrointestinal disorders) | 16 (64)
palmar-plantar erythrodysesthesia (PPES) (Skin and subcutaneous tissue disorders) | 16 (56)
Diarrhea (Gastrointestinal disorders) | 11 (31)
Hypertension (Vascular disorders) | 11 (23)
Mucositis (Gastrointestinal disorders) | 10 (12)
Dysgeusia (Nervous system disorders) | 7 (12)
Anorexia (Metabolism and nutrition disorders) | 5 (11)
Thrombocytopenia (Investigations) | 6 (52) — Platelet count decreased
AST/ALT increased (Investigations) | 3 (11)
Anemia (Blood and lymphatic system disorders) | 3 (15)
Hypothyroidism (Endocrine disorders) | 3 (4)
Neutropenia (Investigations) | 3 (31) — Neutrophil count decreased

LIMITATIONS AND CAVEATS:
Some patients did not have genetic testing and this trial is not able to define prognostic or predictive biomarkers due to small numbers; genetic panel testing varied between institutions and during study period; plasma metanephrine analysis not performed throughout study; only total and not fractionated urinary metanephrines were available; incomplete biochemical interpretation; some standard practices now were not integrated when study initiated in May 2009

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT00843037/Prot_SAP_000.pdf